CLINICAL TRIAL: NCT04116697
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Acupuncture Versus Aromatherapy as Treatments to Lessen Nausea, Vomiting and Anxiety Associated With Adriamycin and Cytoxan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-19-773
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2022-07

CONDITIONS: Nausea; Vomiting; Anxiety
MeSH Terms: conditions — Nausea; Vomiting; Anxiety Disorders | interventions — Acupuncture Therapy; Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupuncture with Anti-Emetics (Experimental)
  Interventions: Other: Acupuncture
- Aromatherapy with Anti-Emetics (Experimental)
  Interventions: Other: Aromatherapy
- Control Group (No Intervention)

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a form of alternative medicine in which thin needles are inserted into the body.
  Arms: Acupuncture with Anti-Emetics
Other: Aromatherapy — Aromatherapy is a form of alternative medicine in which you will inhale aromatic plant extracts and essential oils.
  Arms: Aromatherapy with Anti-Emetics

SUMMARY:
The overall goal of this study is to explore the effectiveness of using acupuncture versus aromatherapy, in conjunction with standard of care anti-emetics, to decrease chemotherapy induced nausea, vomiting, and anxiety in breast cancer patients undergoing Adriamycin and Cytoxan. This study also aims to determine if aromatherapy and anti-emetics is more effective than acupuncture and anti-emetics in treating nausea, vomiting, and anxiety in patients receiving Adriamycin and Cytoxan and if acupuncture and anti-emetics is more effective than aromatherapy and anti-emetics in treating nausea, vomiting, and anxiety in patients receiving Adriamycin and Cytoxan.

ELIGIBILITY:
i) Inclusion

* At least 18 years of age on the day of signing informed consent
* Patient has a diagnosis of breast cancer
* Patient is planned to start Adriamycin and Cytoxan chemotherapy

ii) Exclusion

* Patients who are unable to adhere to the protocol or treatment schedule
* Patients who have a concurrent illness or take medication that induces nausea independent of chemotherapy
* Patients undergoing radiotherapy or hormone therapy during chemotherapy treatments
* Patients who have a sensitive and/or poor sense of smell
* Patients who are allergic to essential oils, specifically peppermint, ginger, and/or lavender
* Patients who are already using essential oils or acupuncture for symptom management and are unwilling to stop while participating in this study
* Patients who are afraid of or unwilling to receive acupuncture stimulation
* Patients who are allergic to stainless steel needles
* Thrombocytopenia (Platelets < 20,000)
* Patients who have received aromatherapy and/or acupuncture treatment within 1 week of starting treatment on this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Nausea | 45 days
  Patients will complete an Edmonton Symptom Assessment Scale. Patients will rate their level of nausea from 0-10 with 10 being the worst possible nausea. Patients will also complete a symptom diary where they will track their level of nausea and how often they are nauseous. Patients will also complete an Anti-Emetic Diary which will track how often they are taking their anti-emetic medications to combat nausea.
improvement in anxiety | 45 days
  Patients will complete an Edmonton Symptom Assessment Scale. Patients will rate their level of anxiety from 0-10 with 10 being the worst possible anxiety. Patients will also complete a symptom diary where they will track their level of anxiety and how often they are anxious.
improvement in vomiting | 45 days
  Patients will complete a symptom diary where they will track how often they vomit. Patients will also complete an Anti-Emetic Diary which will track how often they are taking their anti-emetic medications to combat vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Health, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No